CLINICAL TRIAL: NCT05092464
Title: An Open-Labeled Exploratory Study to Evaluate the Application of Natural Lactic Acid-enriched Cream in Adults With Atopic Dermatitis
Brief Title: Exploratory Study to Evaluate the Application of NLAC Cream in Adults With Atopic Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLACCLAS01
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Staphylococcus Aureus; Atopic Dermatitis
MeSH Terms: conditions — Staphylococcal Infections; Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm open label study (Experimental): 12 week-treatment of 5% natural lactic acid-enriched cream (BID)
  Interventions: Device: Natural Lactic Acid-enriched Cream

INTERVENTIONS:
Device: Natural Lactic Acid-enriched Cream — The subjects were required to topically apply natural lactic acid-enriched cream twice daily in the morning and evening for the treatment duration of 12 weeks.

SUMMARY:
Atopic dermatitis (AD) is the most common chronic inflammatory skin disorder, with a lifetime prevalence of 15-25% in children and 1-3% in adults worldwide. AD is a heterogeneous disease induced by multiple factors, including genetic mutation and environmental risk factors. The main inflammatory mechanism that contributed to AD is the immune response mediated by T helper 2 (Th2) cells. The clinical features of AD, such as recurrent eczematous lesions, IgE-mediated intense itch, and the disruption of skin barrier induced by abnormal epidermal cell differentiation and protein structures, etc., can be attributed to the secretion of Th2 cell-related cytokines. AD is likely to be a lifelong illness with repeated onsets, causing not only physiological discomfort but also psychological distress; hence the quality of life of AD patients is inevitably affected.

Lactic acid is a natural moisturizing factor, which exists in healthy skin. It can efficiently prevent water loss from the skin and alleviate allergic reactions caused by dry skin. The moisturized function of lactic acid has made it became a commonly used additive in a wide variety of skincare products, such as lotion, cream, butter and spray. This product is rich in natural lactic acid generated by the fermentation of probiotics, and therefore can relieve skin itching caused by skin dryness, and resume the water-holding capability of the skin by removing abnormally proliferative stratum corneum as well as inducing collagen production. Importantly, this product is a steroid-free product with safety and without any induced adverse effects in use. This product is also can be a promising option other than steroids to be applied for the mitigation of recurrent symptoms in atopic dermatitis by resuming the water-retention ability of skin and rebuilding skin barrier function.

DETAILED DESCRIPTION:
I. Study Purpose

* Hypothesis:

Natural lactic acid-enriched cream improves the Eczema Area and Severity Index scores in AD patients through inhibiting S. aureus colonization.

- Primary Objective: The primary objective of this study is to assess the clinical efficacy of natural lactic acid-enriched cream for the improvement of Eczema Area and Severity Index (EASI) score in patients with atopic dermatitis.

* Secondary Objectives:

  1. To assess the safety of 12 week-treatment of natural lactic acid-enriched cream, as determined by the count of serious and non-serious treatment-emergent adverse events (AEs) during the time period of every week per participant within each group.
  2. To evaluate the clinical efficacy of natural lactic acid-enriched cream in subjects with atopic dermatitis by Eczema Area and Severity Index (EASI).
  3. To evaluate the clinical efficacy of natural lactic acid-enriched cream in subjects with atopic dermatitis by SCORing Atopic Dermatitis (SCORAD).
  4. To evaluate the clinical efficacy of natural lactic acid-enriched cream in subjects with atopic dermatitis by Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD).
  5. To evaluate the clinical efficacy of natural lactic acid-enriched cream in subjects with atopic dermatitis by Pruritus Numerical Rating Scale (NRS).
  6. To evaluate the clinical efficacy of natural lactic acid-enriched cream in subjects with atopic dermatitis by Trans-epidermal Water Loss (TWEL).
* Exploratory Objectives:

  1. To identify the diversity of the skin microbiome by DNA sequencing at day1 baseline visit, weeks 4, 12 and 16 of natural lactic acid-enriched cream.
  2. To compare the effect of 12 weeks of natural lactic acid-enriched cream treatment on S. aureus abundance for up to 4 weeks after completion of treatment.
  3. To compare the change of S. aureus abundance at day1 baseline visit, weeks 4, 12 and 16 of natural lactic acid-enriched cream application.

     II. Study Design and Methodology

  1. Subject This is a one-arm exploratory trial to evaluate the efficacy and safety of topical application of natural lactic acid-enriched cream on atopic dermatitis. Patients with atopic dermatitis in the ages of 12 to 65 years, with body surface area between 10% and 20% and an Investigator's Global Assessment score of 3 ( moderate) at baseline, will be enrolled in this study.
* Sample size:

Approximately 10 subjects who meet the criteria for study enrollment, will be treated with natural lactic acid-enriched cream.

- Treatment duration: The subjects were required to topically apply natural lactic acid-enriched cream twice daily in the morning and evening for the treatment duration of 12 weeks.

The study includes 3 periods: screening (up to 4 weeks), treatment (12 weeks), and post-treatment follow-up (4 weeks). Study visits occur at screening; at weeks 1, 2, 4, 8 and 12; and 2 and 4 weeks after the completion of treatment (weeks 14 and 16). The study will be conducted in the Department of Dermatology, Taipei Medical School-Shuang Ho Hospital, Ministry of Health and Welfare.

* Inclusion Criteria:

  1. The subject is male or female between 12 and 65 years of age. 2. The subject has a physician-confirmed diagnosis of chronic atopic dermatitis according to Hanifin and Rajka criteria and having active inflammation.

  3. Body surface area (BSA) involvement between 10% and 20%, excluding scalp, at baseline.

  4. An IGA of atopic dermatitis score of 3 at baseline. 5. At least one target lesion that measure at least 3 centimeter (cm) x 3 cm in size at Screening and Baseline and must be representative of the subject's disease state, but not located on the hands, feet, or genitalia.
* Exclusion Criteria:

  1. Unstable course of atopic dermatitis (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks prior to Baseline.
  2. Used any of the following treatments within the indicated washout period before the baseline visit: 12 weeks or 5 half-lives (whichever is longer) - biologic agents (eg, 18 weeks for omalizumab); 8 weeks - cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg, mycophenolate or tacrolimus); 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs; 1 weeks - topical treatments: corticosteroids, calcineurin inhibitors, or coal tar (on the body); 2 weeks - sedating antihistamines (non sedating antihistamines are permitted); 1 week - topical antibiotics, antibacterial cleansing body wash/soap or diluted sodium hypochlorite "bleach" baths.
  3. Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 4 weeks prior to the baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the subject's atopic dermatitis.
  4. The subject planned or anticipated use of any prohibited medications and procedures during study treatment.
  5. Active bacterial, viral, or fungal skin infections.
  6. Participants with any systemic disorder, active skin disease or subjects who present with scars, moles, tattoos, sunburn in the test area which could interfere with the assessment of lesions at screening.
  7. Participant who is immunocompromised (e.g. history of lymphoma, Human Immunodeficiency Virus (HIV)/ Acquired Immune Deficiency Syndrome (AIDS), Wiskott-Aldrich Syndrome) or has a history of malignant disease (with the exception of non- melanoma skin cancer).
  8. Participants with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol.
  9. Subjects have an allergic history of soybean and soybean-derivatives.
  10. Pregnant or lactating females, or females who desire to become pregnant and/or breast feed within the duration of study participation.
  11. The subject planned or anticipated major surgical procedure during the patient's participation in this study.
* Primary Endpoint:

The mean change from baseline in EASI at week 12.

* Secondary Endpoints:

  1. The occurrence of at least one serious or non-serious treatment-emergent AE during the time period of day1 to week 12.
  2. Proportion of patients with EASI 75 ( ≥75% improvement from baseline) at weeks 1, 2, 4, 8, 12, 14 and 16.
  3. The mean percentage change from baseline in EASI score at weeks 1, 2, 4, 8, 12, 14 and 16.
  4. Proportion of patients with both vIGA-AD 0 to 1and a reduction from baseline of ≥2 points at weeks 1, 2, 4, 8, 12, 14 and 16.
  5. The mean percentage change from baseline in vIGA-AD score at weeks 1, 2, 4, 8, 12, 14 and 16.
  6. The mean percentage change from baseline in SCORAD score at weeks 1, 2, 4, 8, 12, 14 and 16.
  7. The mean percentage change from baseline in NRS score at weeks 1, 2, 4, 8, 12, 14 and 16.
  8. The mean percenage change from baseline in transepidermal water loss (TEWL)at weeks 1, 2, 4, 8, 12, 14 and 16.
* Safety Endpoint:

  1. The incidence of adverse events.
  2. Experimental Groups: single-arm, natural lactic acid-enriched cream
  3. Clinical sample collection: To explore the diversity of the skin microbiome, skin microbiota will be harvested by swapping method at day 1 baseline visit, weeks 4, 12 and 16. DNA sequencing will be applied to clarify the composition of cutaneous microbiota at indicated time points.

     III. Statistical Analysis
* General Statistics:

For continuous variables, the following will be presented: mean, median, standard deviation, minimum and maximum. The comparison between two treatment groups and the comparison within group will be tested by using two independent t-test and paired t-test, respectively. If the normal assumption is violated, the Wilcoxon rank-sum and Wilcoxon signed-rank test will be conducted, respectively.

For categorical variables, the numbers and percentages of subjects will be listed and summarized. Comparison for percentages will be performed using the Chi-square test and McNemar's test when comparing results in the same patient. The Fisher's exact test will replace the Chi-square test when any counting of the expected frequency is less than 5.

- Endpoints: To perform the primary efficacy and other endpoints for continuous variable, two independent t-test will be used. If the normal assumption is violated, the non-parametric method of Wilcoxon rank-sum test will be applied for analysis. Significant level will be adopted with two-side at 0.05.

For categorical variables, the Chi-square test will be used. When any counting of the expected frequency is less than 5, the Fisher's exact test will be conducted. Significant alpha level will be adopted at 0.05

- Safety: Adverse events will be coded by preferred term (PT) and system organ class (SOC) by the latest version of MedDRA. Adverse events will be summarized by severity, relationship to study drug, SAEs, and AEs leading to discontinuation of study drug.

Physical examination findings will be presented in a tabulated listing.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female between 12 and 65 years of age.
2. The subject has a physician-confirmed diagnosis of chronic atopic dermatitis according to Hanifin and Rajka criteria and having active inflammation.
3. Body surface area (BSA) involvement between 10% and 20%, excluding scalp, at baseline.
4. An IGA of atopic dermatitis score of 3 at baseline.
5. At least one target lesion that measure at least 3 centimeter (cm) x 3 cm in size at Screening and Baseline and must be representative of the subject's disease state, but not located on the hands, feet, or genitalia.

Exclusion Criteria:

1. Unstable course of atopic dermatitis (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks prior to Baseline.
2. Used any of the following treatments within the indicated washout period before the baseline visit: 12 weeks or 5 half-lives (whichever is longer) - biologic agents (eg, 18 weeks for omalizumab); 8 weeks - cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg, mycophenolate or tacrolimus); 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs; 1 weeks - topical treatments: corticosteroids, calcineurin inhibitors, or coal tar (on the body); 2 weeks - sedating antihistamines (non sedating antihistamines are permitted); 1 week - topical antibiotics, antibacterial cleansing body wash/soap or diluted sodium hypochlorite "bleach" baths.
3. Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 4 weeks prior to the baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the subject's atopic dermatitis.
4. The subject planned or anticipated use of any prohibited medications and procedures during study treatment.
5. Active bacterial, viral, or fungal skin infections.
6. Participants with any systemic disorder, active skin disease or subjects who present with scars, moles, tattoos, sunburn in the test area which could interfere with the assessment of lesions at screening.
7. Participant who is immunocompromised (e.g. history of lymphoma, Human Immunodeficiency Virus (HIV)/ Acquired Immune Deficiency Syndrome (AIDS), Wiskott-Aldrich Syndrome) or has a history of malignant disease (with the exception of non- melanoma skin cancer).
8. Participants with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol.
9. Subjects have an allergic history of soybean and soybean-derivatives.
10. Pregnant or lactating females, or females who desire to become pregnant and/or breast feed within the duration of study participation.
11. The subject planned or anticipated major surgical procedure during the patient's participation in this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
EASI | Week 12
  The mean change from baseline in EASI at week 12.